CLINICAL TRIAL: NCT01246648
Title: Chronic Presence of Epstein Barr Virus in Sulcular and Junctional Epithelial Tissue From Gingiva is Associated With Severe Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 10-PP-13
Record Dates: First submitted 2010-11-17; First posted 2010-11-23 (Estimated); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Parodontitis Aggressive; Parodontitis Chronic
MeSH Terms: interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- chronic periodontitis (Active Comparator)
  Interventions: Procedure: Biopsy
- agressive periodontitis (Active Comparator)
  Interventions: Procedure: biopsy
- healthy patients (Active Comparator)
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — dental extraction and gingival epithelial biopsy
  Arms: chronic periodontitis
Procedure: biopsy — dental extraction and gingival epithelial biopsy
  Arms: agressive periodontitis
Procedure: Biopsy — dental extraction and gingival epithelial biopsy
  Arms: healthy patients

SUMMARY:
The etiopathogenesis of periodontal disease results from complex interaction between infectious agents, mainly including bacteria, and host cellular and humoral immune responses. However it is thought that bacteria-induced pathogenesis is not sufficient alone to explain all biological and clinical features of the destructive periodontal disease. The main hypothesis is that herpesviruses, such as Epstein-Barr Virus, may participate as well by altering epithelial gingival cell biology and consequently may promote the initiation and progression of periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* Men exclusively
* 12 years minimum
* 2 patients affected by chronic periodontitis
* 2 patients affected by aggressive periodontitis
* 2 healthy patients (orthodontics extraction)
* Subject who have read and understood the information note relative under investigation and who have signed the informed consent
* Subject whose legal representative signed the parental consent (if minor patient)

Exclusion Criteria:

* Patient with contre-indication to dental extraction
* Patient witn serious blood disease
* Patient who exhibits systemic condition incompatible with the realization of the study
* Patient treated with oral retinoids, bisphosphonates, oral anticoagulants and anticonvulsivants
* Patient who presents za buccal carcinoma treated with radiotherapy
* Patient who have received during the past 6 months: anti-inflammatory drugs, anti-cancerous or immunosuppressive chemiotherapy
* Patient who presents a linguistic or psychic incapacity to understand information
* Female patient

Min Age: 12 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-01-17 (Actual); Primary Completion 2015-04-01 (Actual); Study Completion 2015-04-01 (Actual)

PRIMARY OUTCOMES:
Presence/absence of EBV in the epithelial cells of periodontal pockets (by Immunofluorescence and in situ Hybridization | at time = 0 (baseline)

SECONDARY OUTCOMES:
Presence/ absence of latency and/or lytic proteins (by immunofluorescence and in situ hybridization | at time = 0 (baseline)
- Epithelial tissue infected (by Immunofluorescence and In situ Hybridization) : detection of oral gingival epithelium, sulcular epithelium, junctional epithelium. | at time = 0 (baseline)

CONTACTS AND LOCATIONS:
Overall Officials: VINCENT Severine, PH, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Hôpital Saint Roch, Nice, France